CLINICAL TRIAL: NCT07218835
Title: Compact Auto-Aligning Multi -Modal Eye Imaging
Brief Title: Compact Auto-Aligning Multi-Modal Eye Imaging to Diagnose Traumatic Eye Injury
Status: Not yet recruiting | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00117676; HT9425-24-1-0870 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2025-10-16; First posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Ocular Pathologies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Tri-Modality, auto-aligning ocular imaging with compact handheld instrument: Color photography, anterior and posterior segment OCT images with the investigational eye imaging system will be taken of consented participant's eyes presenting within Duke Eye Center and Duke University emergency room
  Interventions: Device: Auto-aligning Ocular imaging instrument

INTERVENTIONS:
Device: Auto-aligning Ocular imaging instrument — Develop a tri-modality, auto-aligning ocular imaging instrument incorporating gross color photography, anterior and posterior segment OCT in a compact, handheld form factor.

SUMMARY:
The purpose of this study is to test an investigational eye imaging device by taking pictures of participants eyes with a single image capture that takes only seconds.

ELIGIBILITY:
Inclusion Criteria:

* Ocular complaints potentially indicating anterior segment pathology (e.g., corneal abrasions, corneal edema, corneal scars)
* Ocular complaints potentially indicating posterior segment pathology (e.g., macular edema, neovascular, macular degeneration)

Exclusion Criteria:

* Participant is unable to be imaged for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Duke Eye Center patients will be drawn from the Eye Center clinics and from Duke Emergency Department consulted by ophthalmologist in the Emergency Department.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants who found the eye imaging device easy to use | up to 2 years
Number of participants who found the eye imaging device mobile | up to 2 years
Number of participants who found the eye imaging device reliable | up to 2 years
Image quality as measured by the number of eye condition diagnoses that match official diagnoses | up to 2 years
  Diagnoses made from the eye imaging device will be compared to the official diagnoses the patients received from a full eye exam in the clinic or emergency department.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Kuo, MD, Principal Investigator — Duke University
Locations (1):
- Duke Eye Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No